CLINICAL TRIAL: NCT06107933
Title: Developmental Impacts of MicroPLastics Exposure in Early Life
Acronym: DIMPLE
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Emory University (Other); Sonoma Technology, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00030652; 23-0314 (Other: UC Boulder)
Record Dates: First submitted 2023-10-03; First posted 2023-10-30 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Infant Development; Breast Feeding; Environmental Exposure
Keywords: microplastic; breastmilk; infant microplastic exposure; gut microbiome; fecal metabolome
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — maternal venous blood samples maternal breastmilk samples maternal stool samples infant stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- City Mother-Infant Pairs: Mother-infant pairs living in a Baltimore City, Maryland zip code exposed to micro and nano plastics.
  Interventions: Other: Observational only
- County Mother-Infant Pairs: Mother-infant pairs living in a Baltimore County, Maryland zip code exposed to micro and nano plastics.
  Interventions: Other: Observational only

INTERVENTIONS:
Other: Observational only — Exposure to micro and nano plastics

SUMMARY:
The goal of this observational study is to characterize and evaluate micro- and nano-plastic (MNP) exposures among mothers and infants in mother-infant dyads 1 or 3 months postpartum living in Baltimore, Maryland. The main questions it aims to answer are:

* What MNPs are present in breastmilk and maternal blood samples and in their infants stool sample?
* Are there associations between amount of maternal MNPs in breast milk and mass of MNP particles in infant stool?
* Which environmental and lifestyle factors are most predictive of maternal MNP burden?
* Is infant exposure to MNPs associated with birth weight and postnatal growth trajectories?

Participants will:

* Complete several questionnaires assessing medical histories, lifestyle factors, environmental exposures, eating behaviors, etc.
* Provide biological specimens including: maternal blood, stool, and breastmilk; infant stool
* Clinical visit to have anthropometric measures documented including maternal height and weight, infant weight, length, and skin-fold thickness

DETAILED DESCRIPTION:
The proposed pilot study will establish a new cohort of healthy, lactating women from Baltimore City and Baltimore County, Maryland. By recruiting women from these two regions, the investigators will be able to ensure that the pilot study covers a diverse geographical range with varying levels of air pollution exposure and social determinants of health (SDoH). Study participants will be 1 or 3 months postpartum (+/- 2 weeks) and report exclusive breastfeeding. The investigators will also biobank maternal stool samples for future funding applications that will additionally examine the gut microbiome and fecal metabolome.

Height, Weight, Blood Pressure, and other Anthropometric Measures: Maternal height and weight will be measured using a calibrated medical scale and a commercial stadiometer. Infant weight will be measured in duplicate on a digital scale accurate to the nearest 10 g and length will be measured in duplicate to the nearest 0.1 cm using an Infantometer and the standardized World Health Organization (WHO) approach. Infant skinfold thickness will be measured at four sites with Holtain skinfold callipers. Maternal weight will be recorded to the nearest 0.1 kg and height will be recorded to the nearest 0.1 cm. Automated blood pressure using appropriate cuffs will be used to obtain three readings of blood pressure, from which the average value will be recorded, per recommendations of the American Heart Association.

Assessment of Food Intake; Physical Activity: Dietary data will be collected using the National Cancer Institute (NCI) National Health and Nutritional Examination Survey (NHANES) Food Frequency Questionnaire. The questionnaire is designed to capture information about food intake over the prior month, and includes questions outlining consumption of fruits, vegetables, dairy products, whole grain and fiber, sugar, and red and processed meats. The questionnaire will be administered on the web with a research assistant nearby to assist with any questions. Given the investigators are interested in microplastics exposure from food, additional dietary data will be collected through the administration of Nutrition Data System for Research (NDSR) 24-hour dietary recalls which will be administered over the phone by a registered dietician or study staff under the direct supervision of a registered dietician. The investigators will ask mothers to complete 3 dietary recalls for themselves and 3 for their infant, for ideally 2 weekdays and a weekend. One dietary recall for both mother and infant will be completed during the Clinical Visit at the Clinical Research Unit (CRU). Research assistants will work together with participants to establish which days are best suited for them to complete subsequent recalls. Finally, to assess the quantity of milk consumed by infants during a single feeding, the investigators will weigh the infants at the study visit before feeding. Then mothers will be asked to breastfeed their infant. Upon completion of feeding, the investigators will re-weigh the infants to roughly capture the amount of milk consumed.

Maternal and Infant Fecal Samples: Fecal collection kits will be given to eligible participants. To avoid plastic contamination, maternal fecal collection kits will include an absorbent pad covering any plastic on the stool collection hat, gloves, a metal spoon, and glass container. For the infant stool collection, mothers will be provided with a diaper, bee's wrap; cloth, and all collection supplies that are free of plastic. The investigators will deliver these collection supplies and instructions to participants prior to their visit so that participants may collect these samples at home. The investigators will ask them to take the samples within 24 hours of the visit time to preserve the microbial composition of the stool samples. The instructions will specify that samples should be stored in the refrigerator until their visit. The investigators will provide a cooler for participants to transport the samples to the CRU. If for any reason, participants were not able to obtain these samples at home, participants will be allowed to collect them during the visit, If collected at the clinical visit, maternal and infant stool samples will be transferred into 3-4 glass vials and stored in a -4°C fridge for 24 hours prior to being stored at -80°C for MNP and gut microbiome sequencing. Fecal collection tubes utilize a fecal preservative, which prevents changes to aerobic and anaerobic bacteria that can occur during shipment. Fecal sequencing will be performed at Emory University (Dr. Doug Walker). Only de-identified samples will be sent to Dr. Walker's lab. DNA will be sequenced on the Illumina HiSeq 4000 platform. Microbial composition profiles will be predicted using MetaPhlan. Samples will be functionally mapped using HUMAnN2 to obtain abundance level of gene families from the UniProt Reference Clusters that will be further mapped to MetaCyc metabolic pathways database. Genes will be grouped in clusters of orthologous groups from EggNOG data. Gene family abundances will be grouped into broader functional categories based on annotation for the UniProt gene ontology. For the metabolomics analysis, fecal samples will be analyzed using ultra-performance liquid chromatography (UPLC) and high resolution/tandem mass spectrometry (MS/MS) by Metabolon. Compounds of exogenous, human, and microbial origin will be identified by comparison to library entries of purified standards or recurrent unknown entities. Metabolon maintains a reference library of more than 4,500 known metabolites and more than 9,000 novel metabolites. Biochemical identifications will be based on three criteria: retention index, accurate mass match to the library +/- 10 ppm, and the MS/MS forward and reverse scores between the experimental data and authentic standards.

Breast Milk Expression: Due to potential exposures from feeding breast milk from plastic bottles, all mothers will be asked to only feed their infants from the breast for 14 days prior to infant stool collection. Similar to the stool collection supplies, the investigators will provide mothers with a Haakaa Silicone Breast Pump, silicone storage container with cap, and instructions prior to the study visit. Mothers will be asked to provide a full expression of a single breast. If mothers are uncomfortable providing a full expression, study coordinators will work with mothers to determine an amount appropriate for collection. The investigators will collect a minimum of roughly 4g of breast milk. If mothers are unable to collect their breastmilk sample before the visit, mothers will be provided with a quiet, private CRU study room to pump using a Haakaa Silicone Breast Pump into a silicone storage container. Following collection, a member of our study team will aliquot measures into glass sterile tubes for storage. Following collection, all samples will be stored at -80 degrees C prior to processing and analysis.

Blood Draw: Blood draws will be collected (40mL) for microplastics analysis. Blood will be collected using a stainless steel 21G needle that is connected to a glass container under vacuum, so blood drawn directly from participant is deposited in the glass vacutainer. Glass vacutainers will have a rubber seal for storage.

ELIGIBILITY:
Inclusion Criteria:

* All gender expressions
* Mothers at 1 or 3 months postpartum (± 2 weeks)
* Intent to exclusively breastfeed for ≥ 6 months
* Nulliparous and singleton births
* Receiving only breast milk from the mother, with no formula supplementation

Exclusion Criteria:

* Physical, mental, or cognitive disability that prevents participation; current incarceration
* Chronic conditions in mother and/or infant (e.g., heart disease, cancer, autoimmune disease, diabetes, intestinal bowel syndrome/disease), conditions diagnosed for the first time during pregnancy (e.g. gestational diabetes), neurological conditions in mother and/or infant (e.g. epilepsy, seizures), psychological conditions in mother and/or infant (e.g. bipolar disorder), or neurological/psychological conditions diagnosed in mother during or immediately after pregnancy (e.g. postpartum depression)
* Previously diagnosed with any major illness (e.g., intrauterine growth restriction, birth asphyxia, cancer) or eating disorder or previous gastric band surgery
* Maternal antibiotic use during pregnancy or the postpartum period. Infant antibiotic use at any time during life or taking medications that could affect plastic exposure or the microbiome, such as medications administered via a plastic syringe.
* Use of any breast pump except the Silicon Breast Pump for the 14 days prior to the clinical visit.
* PHQ9 score greater than or equal to 10 indicating clinically relevant symptoms of moderate or worse depression
* Infants who are intersex
* Smoking, drug use (including marijuana use), or alcohol abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include 20 mother-infant pairs from Baltimore City and County. We will be studying lactating mothers at 1 or 3 months postpartum ±2 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Microplastic composition in maternal breastmilk | 1 or 3 months +/- 2 weeks postpartum
  MNPs are measured using pyrolysis GC-HRMS using a Frontier Multi-Shot Pyrolyzer with Auto-Shot Sampler interfaced to a Trace 1310 gas chromatography system and Thermo Scientific Q Exactive GC Orbitrap GC-MS/MS.
Microplastic composition in maternal venous blood | 1 or 3 months +/- 2 weeks postpartum
  MNPs are measured using pyrolysis GC-HRMS using a Frontier Multi-Shot Pyrolyzer with Auto-Shot Sampler interfaced to a Trace 1310 gas chromatography system and Thermo Scientific Q Exactive GC Orbitrap GC-MS/MS.
Microplastic composition in infant stool | 1 or 3 months +/- 2 weeks postpartum
  MNPs are measured using pyrolysis GC-HRMS using a Frontier Multi-Shot Pyrolyzer with Auto-Shot Sampler interfaced to a Trace 1310 gas chromatography system and Thermo Scientific Q Exactive GC Orbitrap GC-MS/MS.
Infant weight | 1 or 3 months +/- 2 weeks postpartum
  Infant weight will be measured in duplicate on a digital scale accurate to the nearest 10 g
Infant length | 1 or 3 months +/- 2 weeks postpartum
  Infant length will be measured in duplicate to the nearest 0.1 cm using an Infantometer.
Infant skinfold thickness | 1 or 3 months +/- 2 weeks postpartum
  Infant skinfold thickness will be measured at four sites with Holtain skinfold callipers

SECONDARY OUTCOMES:
Maternal stool microbiome composition | 1 or 3 months +/- 2 weeks postpartum
  Maternal stool will be stored in cryovials at -80C for future metagenomic sequencing to analyze the composition of the gut microbiome.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya L Alderete, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- East Baltimore Pediatric Inpatient and Outpatient Clinical Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Background] Geyer R, Jambeck JR, Law KL. Production, use, and fate of all plastics ever made. Sci Adv. 2017 Jul 19;3(7):e1700782. doi: 10.1126/sciadv.1700782. eCollection 2017 Jul. PMID 28776036
- [Background] Veidis EM, LaBeaud AD, Phillips AA, Barry M. Tackling the Ubiquity of Plastic Waste for Human and Planetary Health. Am J Trop Med Hyg. 2021 Nov 8;106(1):12-14. doi: 10.4269/ajtmh.21-0968. No abstract available. PMID 34749307
- [Background] Usman S, Abdull Razis AF, Shaari K, Azmai MNA, Saad MZ, Mat Isa N, Nazarudin MF. The Burden of Microplastics Pollution and Contending Policies and Regulations. Int J Environ Res Public Health. 2022 Jun 1;19(11):6773. doi: 10.3390/ijerph19116773. PMID 35682361
- [Background] Law KL, Starr N, Siegler TR, Jambeck JR, Mallos NJ, Leonard GH. The United States' contribution of plastic waste to land and ocean. Sci Adv. 2020 Oct 30;6(44):eabd0288. doi: 10.1126/sciadv.abd0288. Print 2020 Oct. PMID 33127684
- [Background] Kannan K, Vimalkumar K. A Review of Human Exposure to Microplastics and Insights Into Microplastics as Obesogens. Front Endocrinol (Lausanne). 2021 Aug 18;12:724989. doi: 10.3389/fendo.2021.724989. eCollection 2021. PMID 34484127
- [Background] Sendra M, Pereiro P, Figueras A, Novoa B. An integrative toxicogenomic analysis of plastic additives. J Hazard Mater. 2021 May 5;409:124975. doi: 10.1016/j.jhazmat.2020.124975. Epub 2020 Dec 26. PMID 33388451
- [Background] Rustagi N, Pradhan SK, Singh R. Public health impact of plastics: An overview. Indian J Occup Environ Med. 2011 Sep;15(3):100-3. doi: 10.4103/0019-5278.93198. PMID 22412286
- [Background] Yang H, He Y, Yan Y, Junaid M, Wang J. Characteristics, Toxic Effects, and Analytical Methods of Microplastics in the Atmosphere. Nanomaterials (Basel). 2021 Oct 17;11(10):2747. doi: 10.3390/nano11102747. PMID 34685192
- [Background] Yong CQY, Valiyaveettil S, Tang BL. Toxicity of Microplastics and Nanoplastics in Mammalian Systems. Int J Environ Res Public Health. 2020 Feb 26;17(5):1509. doi: 10.3390/ijerph17051509. PMID 32111046
- [Background] Leslie HA, van Velzen MJM, Brandsma SH, Vethaak AD, Garcia-Vallejo JJ, Lamoree MH. Discovery and quantification of plastic particle pollution in human blood. Environ Int. 2022 May;163:107199. doi: 10.1016/j.envint.2022.107199. Epub 2022 Mar 24. PMID 35367073
- [Background] Luqman A, Nugrahapraja H, Wahyuono RA, et al. Microplastic Contamination in Human Stools, Foods, and Drinking Water Associated with Indonesian Coastal Population. Environments. 2021;8(12):138. doi:10.3390/environments8120138
- [Background] Zhang N, Li YB, He HR, Zhang JF, Ma GS. You are what you eat: Microplastics in the feces of young men living in Beijing. Sci Total Environ. 2021 May 1;767:144345. doi: 10.1016/j.scitotenv.2020.144345. Epub 2020 Dec 31. PMID 33434834
- [Background] Schwabl P, Koppel S, Konigshofer P, Bucsics T, Trauner M, Reiberger T, Liebmann B. Detection of Various Microplastics in Human Stool: A Prospective Case Series. Ann Intern Med. 2019 Oct 1;171(7):453-457. doi: 10.7326/M19-0618. Epub 2019 Sep 3. PMID 31476765
- [Background] Yan Z, Liu Y, Zhang T, Zhang F, Ren H, Zhang Y. Analysis of Microplastics in Human Feces Reveals a Correlation between Fecal Microplastics and Inflammatory Bowel Disease Status. Environ Sci Technol. 2022 Jan 4;56(1):414-421. doi: 10.1021/acs.est.1c03924. Epub 2021 Dec 22. PMID 34935363
- [Background] Liu S, Guo J, Liu X, Yang R, Wang H, Sun Y, Chen B, Dong R. Detection of various microplastics in placentas, meconium, infant feces, breastmilk and infant formula: A pilot prospective study. Sci Total Environ. 2023 Jan 1;854:158699. doi: 10.1016/j.scitotenv.2022.158699. Epub 2022 Sep 13. PMID 36108868
- [Background] Zhang J, Wang L, Kannan K. Polyethylene Terephthalate and Polycarbonate Microplastics in Pet Food and Feces from the United States. Environ Sci Technol. 2019 Oct 15;53(20):12035-12042. doi: 10.1021/acs.est.9b03912. Epub 2019 Sep 26. PMID 31525038
- [Background] Ragusa A, Svelato A, Santacroce C, Catalano P, Notarstefano V, Carnevali O, Papa F, Rongioletti MCA, Baiocco F, Draghi S, D'Amore E, Rinaldo D, Matta M, Giorgini E. Plasticenta: First evidence of microplastics in human placenta. Environ Int. 2021 Jan;146:106274. doi: 10.1016/j.envint.2020.106274. Epub 2020 Dec 2. PMID 33395930
- [Background] Zhu L, Zhu J, Zuo R, Xu Q, Qian Y, An L. Identification of microplastics in human placenta using laser direct infrared spectroscopy. Sci Total Environ. 2023 Jan 15;856(Pt 1):159060. doi: 10.1016/j.scitotenv.2022.159060. Epub 2022 Sep 26. PMID 36174702
- [Background] Jenner LC, Rotchell JM, Bennett RT, Cowen M, Tentzeris V, Sadofsky LR. Detection of microplastics in human lung tissue using muFTIR spectroscopy. Sci Total Environ. 2022 Jul 20;831:154907. doi: 10.1016/j.scitotenv.2022.154907. Epub 2022 Mar 29. PMID 35364151
- [Background] Pauly JL, Stegmeier SJ, Allaart HA, Cheney RT, Zhang PJ, Mayer AG, Streck RJ. Inhaled cellulosic and plastic fibers found in human lung tissue. Cancer Epidemiol Biomarkers Prev. 1998 May;7(5):419-28. PMID 9610792
- [Background] Ragusa A, Notarstefano V, Svelato A, Belloni A, Gioacchini G, Blondeel C, Zucchelli E, De Luca C, D'Avino S, Gulotta A, Carnevali O, Giorgini E. Raman Microspectroscopy Detection and Characterisation of Microplastics in Human Breastmilk. Polymers (Basel). 2022 Jun 30;14(13):2700. doi: 10.3390/polym14132700. PMID 35808745
- [Background] Ibrahim YS, Tuan Anuar S, Azmi AA, Wan Mohd Khalik WMA, Lehata S, Hamzah SR, Ismail D, Ma ZF, Dzulkarnaen A, Zakaria Z, Mustaffa N, Tuan Sharif SE, Lee YY. Detection of microplastics in human colectomy specimens. JGH Open. 2020 Nov 21;5(1):116-121. doi: 10.1002/jgh3.12457. eCollection 2021 Jan. PMID 33490620
- [Background] Zhang YX, Wang M, Yang L, Pan K, Miao AJ. Bioaccumulation of differently-sized polystyrene nanoplastics by human lung and intestine cells. J Hazard Mater. 2022 Oct 5;439:129585. doi: 10.1016/j.jhazmat.2022.129585. Epub 2022 Jul 12. PMID 35850063
- [Background] Senathirajah K, Attwood S, Bhagwat G, Carbery M, Wilson S, Palanisami T. Estimation of the mass of microplastics ingested - A pivotal first step towards human health risk assessment. J Hazard Mater. 2021 Feb 15;404(Pt B):124004. doi: 10.1016/j.jhazmat.2020.124004. Epub 2020 Oct 6. PMID 33130380
- [Background] Hirt N, Body-Malapel M. Immunotoxicity and intestinal effects of nano- and microplastics: a review of the literature. Part Fibre Toxicol. 2020 Nov 12;17(1):57. doi: 10.1186/s12989-020-00387-7. PMID 33183327
- [Background] Campanale C, Massarelli C, Savino I, Locaputo V, Uricchio VF. A Detailed Review Study on Potential Effects of Microplastics and Additives of Concern on Human Health. Int J Environ Res Public Health. 2020 Feb 13;17(4):1212. doi: 10.3390/ijerph17041212. PMID 32069998
- [Background] Pironti C, Ricciardi M, Motta O, Miele Y, Proto A, Montano L. Microplastics in the Environment: Intake through the Food Web, Human Exposure and Toxicological Effects. Toxics. 2021 Sep 16;9(9):224. doi: 10.3390/toxics9090224. PMID 34564375
- [Background] Ivleva NP. Chemical Analysis of Microplastics and Nanoplastics: Challenges, Advanced Methods, and Perspectives. Chem Rev. 2021 Oct 13;121(19):11886-11936. doi: 10.1021/acs.chemrev.1c00178. Epub 2021 Aug 26. PMID 34436873
- [Background] Gasperi J, Wright SL, Dris R, et al. Microplastics in air: Are we breathing it in? Current Opinion in Environmental Science & Health. 2018;1:1-5. doi:10.1016/j.coesh.2017.10.002
- [Background] Cai L, Wang J, Peng J, Tan Z, Zhan Z, Tan X, Chen Q. Characteristic of microplastics in the atmospheric fallout from Dongguan city, China: preliminary research and first evidence. Environ Sci Pollut Res Int. 2017 Nov;24(32):24928-24935. doi: 10.1007/s11356-017-0116-x. Epub 2017 Sep 16. PMID 28918553
- [Background] Zhu X, Huang W, Fang M, Liao Z, Wang Y, Xu L, Mu Q, Shi C, Lu C, Deng H, Dahlgren R, Shang X. Airborne Microplastic Concentrations in Five Megacities of Northern and Southeast China. Environ Sci Technol. 2021 Oct 5;55(19):12871-12881. doi: 10.1021/acs.est.1c03618. Epub 2021 Sep 24. PMID 34559513
- [Background] Klein M, Fischer EK. Microplastic abundance in atmospheric deposition within the Metropolitan area of Hamburg, Germany. Sci Total Environ. 2019 Oct 1;685:96-103. doi: 10.1016/j.scitotenv.2019.05.405. Epub 2019 May 29. PMID 31174127
- [Background] Dehghani S, Moore F, Akhbarizadeh R. Microplastic pollution in deposited urban dust, Tehran metropolis, Iran. Environ Sci Pollut Res Int. 2017 Sep;24(25):20360-20371. doi: 10.1007/s11356-017-9674-1. Epub 2017 Jul 13. PMID 28707239
- [Background] Abbasi S, Keshavarzi B, Moore F, Turner A, Kelly FJ, Dominguez AO, Jaafarzadeh N. Distribution and potential health impacts of microplastics and microrubbers in air and street dusts from Asaluyeh County, Iran. Environ Pollut. 2019 Jan;244:153-164. doi: 10.1016/j.envpol.2018.10.039. Epub 2018 Oct 10. PMID 30326387
- [Background] Dris R, Gasperi J, Saad M, Mirande C, Tassin B. Synthetic fibers in atmospheric fallout: A source of microplastics in the environment? Mar Pollut Bull. 2016 Mar 15;104(1-2):290-3. doi: 10.1016/j.marpolbul.2016.01.006. Epub 2016 Jan 17. PMID 26787549
- [Background] Allen S, Allen D, Phoenix VR, et al. Atmospheric transport and deposition of microplastics in a remote mountain catchment. Nat Geosci. 2019;12(5):339-344. doi:10.1038/s41561-019-0335-5
- [Background] Ambrosini R, Azzoni RS, Pittino F, Diolaiuti G, Franzetti A, Parolini M. First evidence of microplastic contamination in the supraglacial debris of an alpine glacier. Environ Pollut. 2019 Oct;253:297-301. doi: 10.1016/j.envpol.2019.07.005. Epub 2019 Jul 9. PMID 31323612
- [Background] Sridharan S, Kumar M, Singh L, Bolan NS, Saha M. Microplastics as an emerging source of particulate air pollution: A critical review. J Hazard Mater. 2021 Sep 15;418:126245. doi: 10.1016/j.jhazmat.2021.126245. Epub 2021 May 28. PMID 34111744
- [Background] Zhang Y, Kang S, Allen S, Allen D, Gao T, Sillanpää M. Atmospheric microplastics: A review on current status and perspectives. Earth-Science Reviews. 2020;203:103118. doi:10.1016/j.earscirev.2020.103118
- [Background] Prietl B, Meindl C, Roblegg E, Pieber TR, Lanzer G, Frohlich E. Nano-sized and micro-sized polystyrene particles affect phagocyte function. Cell Biol Toxicol. 2014 Feb;30(1):1-16. doi: 10.1007/s10565-013-9265-y. Epub 2013 Nov 29. PMID 24292270
- [Background] Hwang J, Choi D, Han S, Choi J, Hong J. An assessment of the toxicity of polypropylene microplastics in human derived cells. Sci Total Environ. 2019 Sep 20;684:657-669. doi: 10.1016/j.scitotenv.2019.05.071. Epub 2019 May 17. PMID 31158627
- [Background] Xu M, Halimu G, Zhang Q, Song Y, Fu X, Li Y, Li Y, Zhang H. Internalization and toxicity: A preliminary study of effects of nanoplastic particles on human lung epithelial cell. Sci Total Environ. 2019 Dec 1;694:133794. doi: 10.1016/j.scitotenv.2019.133794. Epub 2019 Aug 5. PMID 31756791
- [Background] Weber A, Schwiebs A, Solhaug H, Stenvik J, Nilsen AM, Wagner M, Relja B, Radeke HH. Nanoplastics affect the inflammatory cytokine release by primary human monocytes and dendritic cells. Environ Int. 2022 May;163:107173. doi: 10.1016/j.envint.2022.107173. Epub 2022 Mar 15. PMID 35303527
- [Background] Hahladakis JN, Velis CA, Weber R, Iacovidou E, Purnell P. An overview of chemical additives present in plastics: Migration, release, fate and environmental impact during their use, disposal and recycling. J Hazard Mater. 2018 Feb 15;344:179-199. doi: 10.1016/j.jhazmat.2017.10.014. Epub 2017 Oct 9. PMID 29035713
- [Background] Smith M, Love DC, Rochman CM, Neff RA. Microplastics in Seafood and the Implications for Human Health. Curr Environ Health Rep. 2018 Sep;5(3):375-386. doi: 10.1007/s40572-018-0206-z. PMID 30116998
- [Background] Clemente JC, Ursell LK, Parfrey LW, Knight R. The impact of the gut microbiota on human health: an integrative view. Cell. 2012 Mar 16;148(6):1258-70. doi: 10.1016/j.cell.2012.01.035. PMID 22424233
- [Background] Ogunrinola GA, Oyewale JO, Oshamika OO, Olasehinde GI. The Human Microbiome and Its Impacts on Health. Int J Microbiol. 2020 Jun 12;2020:8045646. doi: 10.1155/2020/8045646. eCollection 2020. PMID 32612660
- [Background] Hills RD Jr, Pontefract BA, Mishcon HR, Black CA, Sutton SC, Theberge CR. Gut Microbiome: Profound Implications for Diet and Disease. Nutrients. 2019 Jul 16;11(7):1613. doi: 10.3390/nu11071613. PMID 31315227
- [Background] Mohajeri MH, Brummer RJM, Rastall RA, Weersma RK, Harmsen HJM, Faas M, Eggersdorfer M. The role of the microbiome for human health: from basic science to clinical applications. Eur J Nutr. 2018 May;57(Suppl 1):1-14. doi: 10.1007/s00394-018-1703-4. PMID 29748817
- [Background] Sun Q, Ren SY, Ni HG. Incidence of microplastics in personal care products: An appreciable part of plastic pollution. Sci Total Environ. 2020 Nov 10;742:140218. doi: 10.1016/j.scitotenv.2020.140218. Epub 2020 Jun 22. PMID 32629242
- [Background] Deng L, Li G, Peng S, Wu J, Che Y. Microplastics in personal care products: Exploring public intention of usage by extending the theory of planned behaviour. Sci Total Environ. 2022 Nov 20;848:157782. doi: 10.1016/j.scitotenv.2022.157782. Epub 2022 Aug 1. PMID 35926605
- [Background] Praveena SM, Shaifuddin SNM, Akizuki S. Exploration of microplastics from personal care and cosmetic products and its estimated emissions to marine environment: An evidence from Malaysia. Mar Pollut Bull. 2018 Nov;136:135-140. doi: 10.1016/j.marpolbul.2018.09.012. Epub 2018 Sep 11. PMID 30509794
- [Background] Lei K, Qiao F, Liu Q, Wei Z, Qi H, Cui S, Yue X, Deng Y, An L. Microplastics releasing from personal care and cosmetic products in China. Mar Pollut Bull. 2017 Oct 15;123(1-2):122-126. doi: 10.1016/j.marpolbul.2017.09.016. Epub 2017 Sep 11. PMID 28911870
- [Background] Cheung PK, Fok L. Evidence of microbeads from personal care product contaminating the sea. Mar Pollut Bull. 2016 Aug 15;109(1):582-585. doi: 10.1016/j.marpolbul.2016.05.046. Epub 2016 May 27. PMID 27237038
- [Background] Anderson AG, Grose J, Pahl S, Thompson RC, Wyles KJ. Microplastics in personal care products: Exploring perceptions of environmentalists, beauticians and students. Mar Pollut Bull. 2016 Dec 15;113(1-2):454-460. doi: 10.1016/j.marpolbul.2016.10.048. Epub 2016 Nov 8. PMID 27836135
- [Background] Luo Y, Gibson CT, Chuah C, Tang Y, Naidu R, Fang C. Raman imaging for the identification of Teflon microplastics and nanoplastics released from non-stick cookware. Sci Total Environ. 2022 Dec 10;851(Pt 2):158293. doi: 10.1016/j.scitotenv.2022.158293. Epub 2022 Aug 27. PMID 36030853
- [Background] Luo Y, Chuah C, Amin MA, Khoshyan A, Gibson CT, Tang Y, Naidu R, Fang C. Assessment of microplastics and nanoplastics released from a chopping board using Raman imaging in combination with three algorithms. J Hazard Mater. 2022 Jun 5;431:128636. doi: 10.1016/j.jhazmat.2022.128636. Epub 2022 Mar 7. PMID 35278972
- [Background] Nawalage NSK, Bellanthudawa BKA. Synthetic polymers in personal care and cosmetics products (PCCPs) as a source of microplastic (MP) pollution. Mar Pollut Bull. 2022 Sep;182:113927. doi: 10.1016/j.marpolbul.2022.113927. Epub 2022 Jul 22. PMID 35878476
- [Background] Rubio-Armendariz C, Alejandro-Vega S, Paz-Montelongo S, Gutierrez-Fernandez AJ, Carrascosa-Iruzubieta CJ, Hardisson-de la Torre A. Microplastics as Emerging Food Contaminants: A Challenge for Food Safety. Int J Environ Res Public Health. 2022 Jan 21;19(3):1174. doi: 10.3390/ijerph19031174. PMID 35162198
- [Background] Kwon JH, Kim JW, Pham TD, Tarafdar A, Hong S, Chun SH, Lee SH, Kang DY, Kim JY, Kim SB, Jung J. Microplastics in Food: A Review on Analytical Methods and Challenges. Int J Environ Res Public Health. 2020 Sep 15;17(18):6710. doi: 10.3390/ijerph17186710. PMID 32942613
- [Background] Zolotova N, Kosyreva A, Dzhalilova D, Fokichev N, Makarova O. Harmful effects of the microplastic pollution on animal health: a literature review. PeerJ. 2022 Jun 14;10:e13503. doi: 10.7717/peerj.13503. eCollection 2022. PMID 35722253
- [Background] Cox KD, Covernton GA, Davies HL, Dower JF, Juanes F, Dudas SE. Human Consumption of Microplastics. Environ Sci Technol. 2019 Jun 18;53(12):7068-7074. doi: 10.1021/acs.est.9b01517. Epub 2019 Jun 5. PMID 31184127
- [Background] Mason SA, Welch VG, Neratko J. Synthetic Polymer Contamination in Bottled Water. Front Chem. 2018 Sep 11;6:407. doi: 10.3389/fchem.2018.00407. eCollection 2018. PMID 30255015
- [Background] Santos AL, Rodrigues CC, Oliveira M, Rocha TL. Microbiome: A forgotten target of environmental micro(nano)plastics? Sci Total Environ. 2022 May 20;822:153628. doi: 10.1016/j.scitotenv.2022.153628. Epub 2022 Feb 3. PMID 35124041
- [Background] Chen G, Feng Q, Wang J. Mini-review of microplastics in the atmosphere and their risks to humans. Sci Total Environ. 2020 Feb 10;703:135504. doi: 10.1016/j.scitotenv.2019.135504. Epub 2019 Nov 13. PMID 31753503
- [Background] Wang Y, Huang J, Zhu F, Zhou S. Airborne Microplastics: A Review on the Occurrence, Migration and Risks to Humans. Bull Environ Contam Toxicol. 2021 Oct;107(4):657-664. doi: 10.1007/s00128-021-03180-0. Epub 2021 Mar 19. PMID 33742221
- [Background] Ferguson L, Taylor J, Davies M, Shrubsole C, Symonds P, Dimitroulopoulou S. Exposure to indoor air pollution across socio-economic groups in high-income countries: A scoping review of the literature and a modelling methodology. Environ Int. 2020 Oct;143:105748. doi: 10.1016/j.envint.2020.105748. Epub 2020 Jul 3. PMID 32629198
- [Background] Islam MM. Social Determinants of Health and Related Inequalities: Confusion and Implications. Front Public Health. 2019 Feb 8;7:11. doi: 10.3389/fpubh.2019.00011. eCollection 2019. No abstract available. PMID 30800646
- [Background] Danopoulos E, Twiddy M, West R, Rotchell JM. A rapid review and meta-regression analyses of the toxicological impacts of microplastic exposure in human cells. J Hazard Mater. 2022 Apr 5;427:127861. doi: 10.1016/j.jhazmat.2021.127861. Epub 2021 Nov 24. PMID 34863566
- [Background] Lear G, Kingsbury JM, Franchini S, Gambarini V, Maday SDM, Wallbank JA, Weaver L, Pantos O. Plastics and the microbiome: impacts and solutions. Environ Microbiome. 2021 Jan 20;16(1):2. doi: 10.1186/s40793-020-00371-w. PMID 33902756
- [Background] Pérez-Guevara F, Roy PD, Kutralam-Muniasamy G, Shruti VC. A central role for fecal matter in the transport of microplastics: An updated analysis of new findings and persisting questions. Journal of Hazardous Materials Advances. 2021;4:100021. doi:10.1016/j.hazadv.2021.100021
- [Background] Biagi E, Musella M, Palladino G, et al. Impact of Plastic Debris on the Gut Microbiota of Caretta caretta From Northwestern Adriatic Sea. Front Mar Sci. 2021;8:637030. doi:10.3389/fmars.2021.637030
- [Background] Zrimec J, Kokina M, Jonasson S, Zorrilla F, Zelezniak A. Plastic-Degrading Potential across the Global Microbiome Correlates with Recent Pollution Trends. mBio. 2021 Oct 26;12(5):e0215521. doi: 10.1128/mBio.02155-21. Epub 2021 Oct 26. PMID 34700384
- [Background] Sanchez C, Franco L, Regal P, Lamas A, Cepeda A, Fente C. Breast Milk: A Source of Functional Compounds with Potential Application in Nutrition and Therapy. Nutrients. 2021 Mar 22;13(3):1026. doi: 10.3390/nu13031026. PMID 33810073
- [Background] Main KM, Mortensen GK, Kaleva MM, Boisen KA, Damgaard IN, Chellakooty M, Schmidt IM, Suomi AM, Virtanen HE, Petersen DV, Andersson AM, Toppari J, Skakkebaek NE. Human breast milk contamination with phthalates and alterations of endogenous reproductive hormones in infants three months of age. Environ Health Perspect. 2006 Feb;114(2):270-6. doi: 10.1289/ehp.8075. PMID 16451866
- [Background] Fromme H, Gruber L, Seckin E, Raab U, Zimmermann S, Kiranoglu M, Schlummer M, Schwegler U, Smolic S, Volkel W; HBMnet. Phthalates and their metabolites in breast milk--results from the Bavarian Monitoring of Breast Milk (BAMBI). Environ Int. 2011 May;37(4):715-22. doi: 10.1016/j.envint.2011.02.008. PMID 21406311
- [Background] Chao HH, Guo CH, Huang CB, Chen PC, Li HC, Hsiung DY, Chou YK. Arsenic, cadmium, lead, and aluminium concentrations in human milk at early stages of lactation. Pediatr Neonatol. 2014 Apr;55(2):127-34. doi: 10.1016/j.pedneo.2013.08.005. Epub 2013 Nov 11. PMID 24231114
- [Background] LaKind JS, Naiman J, Verner MA, Leveque L, Fenton S. Per- and polyfluoroalkyl substances (PFAS) in breast milk and infant formula: A global issue. Environ Res. 2023 Feb 15;219:115042. doi: 10.1016/j.envres.2022.115042. Epub 2022 Dec 16. PMID 36529330
- [Background] Zheng G, Schreder E, Dempsey JC, Uding N, Chu V, Andres G, Sathyanarayana S, Salamova A. Per- and Polyfluoroalkyl Substances (PFAS) in Breast Milk: Concerning Trends for Current-Use PFAS. Environ Sci Technol. 2021 Jun 1;55(11):7510-7520. doi: 10.1021/acs.est.0c06978. Epub 2021 May 13. PMID 33982557
- [Background] LaKind JS, Verner MA, Rogers RD, Goeden H, Naiman DQ, Marchitti SA, Lehmann GM, Hines EP, Fenton SE. Current Breast Milk PFAS Levels in the United States and Canada: After All This Time, Why Don't We Know More? Environ Health Perspect. 2022 Feb;130(2):25002. doi: 10.1289/EHP10359. Epub 2022 Feb 23. PMID 35195447
- [Background] Mielech A, Puscion-Jakubik A, Socha K. Assessment of the Risk of Contamination of Food for Infants and Toddlers. Nutrients. 2021 Jul 9;13(7):2358. doi: 10.3390/nu13072358. PMID 34371868
- [Background] Ljung K, Palm B, Grander M, Vahter M. High concentrations of essential and toxic elements in infant formula and infant foods - A matter of concern. Food Chem. 2011 Aug 1;127(3):943-51. doi: 10.1016/j.foodchem.2011.01.062. Epub 2011 Jan 25. PMID 25214082
- [Background] Balali-Mood M, Naseri K, Tahergorabi Z, Khazdair MR, Sadeghi M. Toxic Mechanisms of Five Heavy Metals: Mercury, Lead, Chromium, Cadmium, and Arsenic. Front Pharmacol. 2021 Apr 13;12:643972. doi: 10.3389/fphar.2021.643972. eCollection 2021. PMID 33927623
- [Background] Chumpitazi B, Nurko S. Pediatric gastrointestinal motility disorders: challenges and a clinical update. Gastroenterol Hepatol (N Y). 2008 Feb;4(2):140-8. PMID 21904491
- [Background] Jadcherla SR, Duong HQ, Hofmann C, Hoffmann R, Shaker R. Characteristics of upper oesophageal sphincter and oesophageal body during maturation in healthy human neonates compared with adults. Neurogastroenterol Motil. 2005 Oct;17(5):663-70. doi: 10.1111/j.1365-2982.2005.00706.x. PMID 16185304
- [Background] Llorca M, Farre M, Pico Y, Teijon ML, Alvarez JG, Barcelo D. Infant exposure of perfluorinated compounds: levels in breast milk and commercial baby food. Environ Int. 2010 Aug;36(6):584-92. doi: 10.1016/j.envint.2010.04.016. Epub 2010 May 21. PMID 20494442
- [Background] Jian JM, Chen D, Han FJ, Guo Y, Zeng L, Lu X, Wang F. A short review on human exposure to and tissue distribution of per- and polyfluoroalkyl substances (PFASs). Sci Total Environ. 2018 Sep 15;636:1058-1069. doi: 10.1016/j.scitotenv.2018.04.380. Epub 2018 May 3. PMID 29913568
- [Background] Cai J, Zang X, Wu Z, Liu J, Wang D. Translocation of transition metal oxide nanoparticles to breast milk and offspring: The necessity of bridging mother-offspring-integration toxicological assessments. Environ Int. 2019 Dec;133(Pt A):105153. doi: 10.1016/j.envint.2019.105153. Epub 2019 Sep 11. PMID 31520958
- [Background] Yang L , Kuang H , Zhang W , Wei H , Xu H . Quantum dots cause acute systemic toxicity in lactating rats and growth restriction of offspring. Nanoscale. 2018 Jun 21;10(24):11564-11577. doi: 10.1039/c8nr01248b. PMID 29892752
- [Background] Yin K, Wang Y, Zhao H, et al. A comparative review of microplastics and nanoplastics: Toxicity hazards on digestive, reproductive and nervous system. Science of The Total Environment. 2021;774:145758. doi:10.1016/j.scitotenv.2021.145758
- [Background] Han Y, Lian F, Xiao Z, Gu S, Cao X, Wang Z, Xing B. Potential toxicity of nanoplastics to fish and aquatic invertebrates: Current understanding, mechanistic interpretation, and meta-analysis. J Hazard Mater. 2022 Apr 5;427:127870. doi: 10.1016/j.jhazmat.2021.127870. Epub 2021 Nov 24. PMID 34848066
- [Background] Liu FF, Liu GZ, Zhu ZL, Wang SC, Zhao FF. Interactions between microplastics and phthalate esters as affected by microplastics characteristics and solution chemistry. Chemosphere. 2019 Jan;214:688-694. doi: 10.1016/j.chemosphere.2018.09.174. Epub 2018 Oct 1. PMID 30292051
- [Background] Hafezi SA, Abdel-Rahman WM. The Endocrine Disruptor Bisphenol A (BPA) Exerts a Wide Range of Effects in Carcinogenesis and Response to Therapy. Curr Mol Pharmacol. 2019;12(3):230-238. doi: 10.2174/1874467212666190306164507. PMID 30848227
- [Background] Peretz J, Vrooman L, Ricke WA, Hunt PA, Ehrlich S, Hauser R, Padmanabhan V, Taylor HS, Swan SH, VandeVoort CA, Flaws JA. Bisphenol a and reproductive health: update of experimental and human evidence, 2007-2013. Environ Health Perspect. 2014 Aug;122(8):775-86. doi: 10.1289/ehp.1307728. Epub 2014 Jun 4. PMID 24896072
- [Background] Rubin BS. Bisphenol A: an endocrine disruptor with widespread exposure and multiple effects. J Steroid Biochem Mol Biol. 2011 Oct;127(1-2):27-34. doi: 10.1016/j.jsbmb.2011.05.002. Epub 2011 May 13. PMID 21605673
- [Background] Henderson NB, Sears CG, Calafat A, et al. Associations of Breast Milk Consumption with Urinary Phthalate and Phenol Exposure Biomarkers in Infants. Environ Sci Technol Lett. 2020;7(10):733-739. doi:10.1021/acs.estlett.0c00450
- [Background] Wick P, Malek A, Manser P, Meili D, Maeder-Althaus X, Diener L, Diener PA, Zisch A, Krug HF, von Mandach U. Barrier capacity of human placenta for nanosized materials. Environ Health Perspect. 2010 Mar;118(3):432-6. doi: 10.1289/ehp.0901200. Epub 2009 Nov 12. PMID 20064770
- [Background] Chambers ES, Preston T, Frost G, Morrison DJ. Role of Gut Microbiota-Generated Short-Chain Fatty Acids in Metabolic and Cardiovascular Health. Curr Nutr Rep. 2018 Dec;7(4):198-206. doi: 10.1007/s13668-018-0248-8. PMID 30264354
- [Background] Lynch CJ, Adams SH. Branched-chain amino acids in metabolic signalling and insulin resistance. Nat Rev Endocrinol. 2014 Dec;10(12):723-36. doi: 10.1038/nrendo.2014.171. Epub 2014 Oct 7. PMID 25287287
- [Background] Defois C, Ratel J, Garrait G, Denis S, Le Goff O, Talvas J, Mosoni P, Engel E, Peyret P. Food Chemicals Disrupt Human Gut Microbiota Activity And Impact Intestinal Homeostasis As Revealed By In Vitro Systems. Sci Rep. 2018 Jul 20;8(1):11006. doi: 10.1038/s41598-018-29376-9. PMID 30030472
- [Background] de la Cuesta-Zuluaga J, Mueller NT, Alvarez-Quintero R, Velasquez-Mejia EP, Sierra JA, Corrales-Agudelo V, Carmona JA, Abad JM, Escobar JS. Higher Fecal Short-Chain Fatty Acid Levels Are Associated with Gut Microbiome Dysbiosis, Obesity, Hypertension and Cardiometabolic Disease Risk Factors. Nutrients. 2018 Dec 27;11(1):51. doi: 10.3390/nu11010051. PMID 30591685
- [Background] Org E, Blum Y, Kasela S, Mehrabian M, Kuusisto J, Kangas AJ, Soininen P, Wang Z, Ala-Korpela M, Hazen SL, Laakso M, Lusis AJ. Relationships between gut microbiota, plasma metabolites, and metabolic syndrome traits in the METSIM cohort. Genome Biol. 2017 Apr 13;18(1):70. doi: 10.1186/s13059-017-1194-2. PMID 28407784
- [Background] Lin H, An Y, Hao F, Wang Y, Tang H. Correlations of Fecal Metabonomic and Microbiomic Changes Induced by High-fat Diet in the Pre-Obesity State. Sci Rep. 2016 Feb 26;6:21618. doi: 10.1038/srep21618. PMID 26916743
- [Background] Wang Lei, Zhang Junjie, Hou Shaogang, Sun Hongwen. A Simple Method for Quantifying Polycarbonate and Polyethylene Terephthalate Microplastics in Environmental Samples by Liquid Chromatography-Tandem Mass Spectrometry. Environmental Science & Technology Letters. 2017;4(12):530-534. doi:10.1021/acs.estlett.7b00454
- [Background] Amtmann D, Kim J, Chung H, Bamer AM, Askew RL, Wu S, Cook KF, Johnson KL. Comparing CESD-10, PHQ-9, and PROMIS depression instruments in individuals with multiple sclerosis. Rehabil Psychol. 2014 May;59(2):220-229. doi: 10.1037/a0035919. Epub 2014 Mar 24. PMID 24661030
- [Background] Andresen EM, Malmgren JA, Carter WB, Patrick DL. Screening for depression in well older adults: evaluation of a short form of the CES-D (Center for Epidemiologic Studies Depression Scale). Am J Prev Med. 1994 Mar-Apr;10(2):77-84. PMID 8037935